CLINICAL TRIAL: NCT06894004
Title: Mechanism of Ketogenic Diet-Induced Hypercholesterolemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202409091
Record Dates: First submitted 2025-03-10; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Hypercholesterolemia and Hyperlipidemia
Keywords: LDL-cholesterol; cholesterol; ketogenic diet; lipoprotein kinetics
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Arm A will complete the Ketogenic Diet intervention first, followed by the Control Diet intervention after a 4-week washout period.
  Interventions: Behavioral: Ketogenic Diet; Behavioral: Control Diet
- B (Experimental): Arm B will complete the Control Diet intervention first, followed by the Ketogenic Diet intervention after a 4-week washout period.
  Interventions: Behavioral: Ketogenic Diet; Behavioral: Control Diet

INTERVENTIONS:
Behavioral: Ketogenic Diet — Participants will consume an isocaloric ketogenic diet for 4 weeks with all food provided as packed-out meals.
Behavioral: Control Diet — Participants will consume an isocaloric control diet for 4 weeks with all food provided as packed-out meals.

SUMMARY:
Very-low carbohydrate ketogenic diets can dramatically increase blood cholesterol levels, particularly in normal-weight people, for reasons that are not well understood. This study will enroll normal-weight adults, will identify "responders" who develop high cholesterol on a ketogenic diet, and will measure rates of production and removal of certain types of cholesterol-carrying particles called lipoproteins in responders. The results will clarify the mechanism by which a ketogenic diet can cause high cholesterol in certain susceptible people.

DETAILED DESCRIPTION:
This study will evaluate the mechanism of ketogenic diet-induced hypercholesterolemia in susceptible normal-weight adults. The first stage of screening will identify eligible young adults who are normal-weight and at low cardiovascular risk. The second stage of screening will identify "responders" who demonstrate susceptibility to ketogenic diet-induced hypercholesterolemia by displaying an increase in LDL-cholesterol concentration after a 3-week screening ketogenic diet. Responders will be eligible to complete a randomized crossover clinical study at Washington University School of Medicine in St. Louis, MO. The randomized crossover study will involve isotope tracer studies of lipoprotein and cholesterol kinetics after two separate 4-week dietary interventions [ketogenic diet and control diet], conducted in random order with a 4-week washout period between interventions. All food will be provided to the participants as packed-out meals. Certain outcomes will use data from the screening process, comparing screen successes and screen failures to evaluate factors that could influence susceptibility to ketogenic diet-induced hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 18 and < 40 years
2. BMI ≥ 18.5 and < 25.0 kg/m2
3. baseline serum LDL-c < 150 mg/dL (< 3.9 mmol/L)
4. baseline serum TG < 100 mg/dL (< 1.1 mmol/L)
5. HbA1c ≤ 5.6%.

Exclusion Criteria:

1. personal or family history of familial hypercholesterolemia
2. current use of lipid-lowering drugs
3. currently on a ketogenic diet and unwilling to change diet
4. current tobacco use
5. hypertension
6. prediabetes or diabetes
7. elevated Lp(a) > 6.5% of ApoB-containing lipoproteins at baseline
8. oral contraceptive use
9. contraindication to heparin
10. known atherosclerotic cardiovascular disease
11. unwilling to abstain from alcohol

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2030-11-30 (Estimated); Study Completion 2030-11-30 (Estimated)

PRIMARY OUTCOMES:
VLDL-ApoB100 production rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and VLDL-ApoB100 leucine isotopic enrichment and compartmental modeling

SECONDARY OUTCOMES:
VLDL-ApoB100 fractional catabolic rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and VLDL-ApoB100 leucine isotopic enrichment and compartmental modeling
IDL-ApoB100 production rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and IDL-ApoB100 leucine isotopic enrichment and compartmental modeling
IDL-ApoB100 fractional catabolic rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and IDL-ApoB100 leucine isotopic enrichment and compartmental modeling
LDL-ApoB100 production rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and LDL-ApoB100 leucine isotopic enrichment and compartmental modeling
LDL-ApoB100 fractional catabolic rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and LDL-ApoB100 leucine isotopic enrichment and compartmental modeling
VLDL-triglyceride production rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and VLDL glycerol isotopic enrichment and compartmental modeling
VLDL-triglyceride fractional catabolic rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and VLDL glycerol isotopic enrichment and compartmental modeling
Plasma lipoprotein lipase activity | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by assaying lipoprotein lipase activity in post-heparin plasma
Plasma lipoprotein profile | At baseline, immediately after the screening ketogenic diet, immediately after the 4-week ketogenic diet intervention period, and immediately after the 4-week control diet intervention period.
  Determined by standard clinical chemistry methods and by advanced lipoprotein profiling
Whole-body lipolytic rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma palmitate isotopic enrichment
Relative contribution of systemic fatty acids to VLDL-triglyceride | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using plasma and VLDL-triglyceride palmitate isotopic enrichment and compartmental modeling
Cholesterol synthetic rate | Immediately after the 4-week ketogenic diet intervention period and immediately after the 4-week control diet intervention period.
  Determined by using mass isotopomer distribution analysis of deuterium enrichment in plasma cholesterol after labeling the total body water pool with deuterium oxide
Fat mass | Immediately after the screening ketogenic diet
  Determined by using dual-energy X-ray absorptiometry
Fat-free mass | Immediately after the screening ketogenic diet
  Determined by using dual-energy X-ray absorptiometry
Insulin sensitivity | Immediately after the screening ketogenic diet
  Determined by measuring fasting plasma glucose, insulin, and C-peptide
Thyroid function | Immediately after the screening ketogenic diet
  Determined by measuring TSH, free T4, and free T3
Adipokines | Immediately after the screening ketogenic diet
  Determined by measuring plasma leptin and adiponectin
Cholesterol absorption markers | Immediately after the screening ketogenic diet
  Determined by measuring serum campesterol, sitosterol, and cholestanol

CONTACTS AND LOCATIONS:
Overall Officials: Max C Petersen, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
All raw data used to generate descriptive statistics presented in manuscripts incorporating results generated from this study will be included as supplemental data files as and when required. Fully de-identified raw data, including all outcome measures and tracer enrichments from kinetic studies will be available in .csv format, which can be manipulated by many free and commercial software packages. Individual-level data will be shared as allowed by informed consent agreements approved by the Institutional Review Board (IRB).
Supporting Information: Study Protocol
Time Frame: Data will be made available upon peer-reviewed publication of the study results or earlier as required by the study sponsor and/or funding sources.
Access Criteria: FAIR Data Sharing protocols will be applied so that the data will be Findable, Accessible, Interoperable, and Re-usable.